CLINICAL TRIAL: NCT04937933
Title: The Effect of Coolant Spray on Rib Fracture Pain of Geriatric Blunt Thoracic Trauma Patients: a Randomized Controlled Trial
Brief Title: Effect of Coolant Spray on Traumatic Rib Pain of Geriatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Abdullah Osman KOCAK, Associate Professor of Emergency Department of Ataturk University, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Ataturk University00001
Record Dates: First submitted 2021-06-17; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Thorax; Fracture; Pain; Thorax, Thoracic, Spine, With Radicular and Visceral Pain
Keywords: Rib fracture; Geriatrics; Coolant Spray; Lidocaine
MeSH Terms: conditions — Fractures, Bone; Pain; Visceral Pain; Rib Fractures | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coolant spray group (Active Comparator): Coolant spray (Cryos ®Spray, Phyto Performance, Italy) was applied as suggested by the manufacturer (at a distance of 20 cm from the injured area for 5-10 s). Saline solution was sprayed for the same duration and at the same distance from the injured area as well. The first spray application was performed after the initial assessment, and the second spray application was performed at the end of the 30th minute (immediately after the pain level/score measurement). All patients were given intravenous (IV) dexketoprofen (50 mg in 50 ml standard saline solution) in 5 minutes simultaneously with the first spray application. The physicians applied the designated treatment protocol for each treatment group. As a rescue analgesic treatment, patients were scheduled to be given IV fentanyl at a dose of 1 mcg/kg.
  Interventions: Drug: Coolant spray (Cryos ®Spray, Phyto Performance, Italy)
- Placebo group (Placebo Comparator): A standard saline solution in a bottle covered with opaque white paper and refrigerated at 4°C was prepared. Saline solution was sprayed for the same duration and at the same distance from the injured area as well like coolant spray application. The first spray application was performed after the initial assessment, and the second spray application was performed at the end of the 30th minute (immediately after the pain level/score measurement). All patients were given intravenous (IV) dexketoprofen (50 mg in 50 ml standard saline solution) in 5 minutes simultaneously with the first spray application. The physicians applied the designated treatment protocol for each treatment group. As a rescue analgesic treatment, patients were scheduled to be given IV fentanyl at a dose of 1 mcg/kg.
  Interventions: Drug: Saline solution

INTERVENTIONS:
Drug: Coolant spray (Cryos ®Spray, Phyto Performance, Italy) — The coolant spray treatment method is a cryotherapy non-pharmacological treatment choice.
  Arms: Coolant spray group
Drug: Saline solution — saline solution
  Arms: Placebo group

SUMMARY:
This study aims to evaluate the effectiveness of cryotherapy in the early period pain treatment of elderly patients with rib fractures due to blunt thoracic trauma.In this prospective randomized controlled study, geriatric patients were assigned to groups to receive either coolant spray (n=51) or placebo spray (n=50). To the coolant spray group patients,a coolant spray was applied. To the placebo group patients, a normal saline solution in a bottle covered with white opaque paper and refrigerated at 4 °C was sprayed. The visual analog scale (VAS) scores of all patients were recorded before starting spray application (V 0 ), at 10th minute (V 1 ), 20th minute (V 2 ), 30th minute (V 3 ), 60th minute (V 4 ), 120th minute (V 5 ), and 360th minute (V 6 ). The mean decreases in the VAS scores and the mean of the percentage of reduction in the VAS scores were calculated.

DETAILED DESCRIPTION:
The study was a prospective, randomized, controlled, double-blind, multicenter clinical trial.All patients were informed about the study procedures, and written consent was obtained from the volunteers, who agreed to participate. Application of the sprays and measurement of the VAS scores were performed by ED physicians who were blinded for the study. For the placebo group, a standard saline solution in a bottle covered with opaque white paper and refrigerated at 4°C was prepared. In the coolant spray group, coolant spray was applied as suggested by the manufacturer (at a distance of 20 cm from the injured area for 5-10 s). Saline solution was sprayed for the same duration and at the same distance from the injured area as well. The first spray application was performed after the initial assessment, and the second spray application was performed at the end of the 30th minute (immediately after the pain level/score measurement). All patients were given intravenous (IV) dexketoprofen (50 mg in 50 ml standard saline solution) in 5 minutes simultaneously with the first spray application. The physicians applied the designated treatment protocol for each treatment group. As a rescue analgesic treatment, patients were scheduled to be given IV fentanyl at a dose of 1 mcg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Trauma developed in less than 24 hours.
* Presence of rib fractures below 3 (6).
* Rib fractures being limited to a single hemithorax.
* Having a visual analog scale (VAS) score of 5 or more.

Exclusion Criteria:

* Inability to provide informed consent (altered mental state, non-Turkish-speaking).
* Patients with chest injury scores above 11 were excluded from the study because of the insufficiency of this multimodal treatment.
* Having additional trauma-related injuries (including lung contusion, pneumothorax, hemothorax, etc.), skin lesions at the site of trauma, and/or trauma-related pain in multiple regions of the thorax.
* Patients with fractures in ribs 1 and 2 (in terms of the risk of serious injury that may accompany).
* History of regular analgesic usage (such as chronic pain syndrome, rheumatoid arthritis, osteoarthritis), antiaggregant and anticoagulant drug usage, and/or allergy to nonsteroidal antiinflammatory drugs (NSAID) and narcotic analgesics.
* History of having coagulation disorders, hematologic disease, gastrointestinal bleeding, uncontrolled heart failure, chronic renal failure, chronic liver failure, and chronic lung disease.
* Patients in whom trauma-related complications developed during the ED follow-up, the general condition worsened, vital signs were unstable, and patients that needed to be hospitalized.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Pain level | 6 hoursa
  The study's primary outcome is determined as a ≥50% reduction (clinical effectiveness) according to the initial VAS score

SECONDARY OUTCOMES:
Rescure Medicine | 6 Hourss
  The secondary outcome variable is the difference between the placebo and coolant spray groups in terms of the frequency of patients that needed at least one dose of rescue treatment during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peek J, Smeeing DPJ, Hietbrink F, Houwert RM, Marsman M, de Jong MB. Comparison of analgesic interventions for traumatic rib fractures: a systematic review and meta-analysis. Eur J Trauma Emerg Surg. 2019 Aug;45(4):597-622. doi: 10.1007/s00068-018-0918-7. Epub 2018 Feb 6. PMID 29411048
- [Background] Gur STA, Dogruyol S, Kocak AO, Akbas I, Tuncer K, Karabulut H, Cakir Z. Comparison of effectiveness coolant spray and placebo in patients with acute ankle trauma prospective randomized controlled trial. Am J Emerg Med. 2020 Jul;38(7):1458-1462. doi: 10.1016/j.ajem.2019.12.054. Epub 2020 Jan 7. PMID 31973934
- [Background] Farion KJ, Splinter KL, Newhook K, Gaboury I, Splinter WM. The effect of vapocoolant spray on pain due to intravenous cannulation in children: a randomized controlled trial. CMAJ. 2008 Jul 1;179(1):31-6. doi: 10.1503/cmaj.070874. PMID 18591524
- [Background] Waterhouse MR, Liu DR, Wang VJ. Cryotherapeutic topical analgesics for pediatric intravenous catheter placement: ice versus vapocoolant spray. Pediatr Emerg Care. 2013 Jan;29(1):8-12. doi: 10.1097/PEC.0b013e31827b214b. PMID 23283254
- [Background] Zhu Y, Peng X, Wang S, Chen W, Liu C, Guo B, Zhao L, Gao Y, Wang K, Lou F. Vapocoolant spray versus placebo spray/no treatment for reducing pain from intravenous cannulation: A meta-analysis of randomized controlled trials. Am J Emerg Med. 2018 Nov;36(11):2085-2092. doi: 10.1016/j.ajem.2018.03.068. Epub 2018 Mar 27. PMID 30253890